CLINICAL TRIAL: NCT03835364
Title: Aptus at Home: Co-design of a Home-based Monitoring System for Anaemia
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS: 233542
Record Dates: First submitted 2018-12-27; First posted 2019-02-08 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Anemia; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Blood measurement — Single fingerprick to measure haemoglobin and haematocrit measurements using the Aptus Home, anaemia home monitoring system.

SUMMARY:
Co-design of a home-based anaemia monitoring system with participants who have previous diagnosis of anaemia.

DETAILED DESCRIPTION:
The device/ monitoring system being developed is called Aptus home. Aptus home measures the haemoglobin and haematocrit levels in blood from a single drop of blood. By measuring these blood parameters, participants are able to monitor anaemia in participants' homes.

The use of the device will take place in the participant's home to simulate what the investigators believe will be the ideal location for people who would prefer to self-manage their condition.

This study is a unique opportunity to gain feedback on the future design and development of a home-based monitoring system through user evaluation. As this is an adaptive/ iterative study design, this will give the Sponsor the opportunity to make changes to the user interface and user platform based on the feedback received from the end user.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of anaemia
* Commitment to perform finger pricking to use the device every two weeks and complete 2 monthly questionnaires
* Participant's willingness to participate in 1 to 1 interviews and, or focus groups
* Understands and has a good level of spoken and written English

Exclusion Criteria:

* No prior diagnosis of anaemia
* Not committed to perform two weekly finger pricks to use device and complete 2 monthly questionnaires
* Unwilling to attend interviews and focus groups
* Doesn't have a good level of written and spoken English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone over 18 years of age with a prior diagnosis of anaemia, who have the capability to sign consent for the themselves and commit to the requirements of the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Qualitative capture of user feedback- Questionnaires | 14 months
  User feedback gathered from participants using the anaemia monitoring device in participants' homes will be used to inform the changes necessary to develop a successful home-based anaemia monitoring system.
Qualitative capture of user feedback- focus groups | 14 months
  User feedback gathered from participants using the anaemia monitoring device in participants' homes will be used to inform the changes necessary to develop a successful home-based anaemia monitoring system.

CONTACTS AND LOCATIONS:
Locations (1):
- Entia Ltd, Room G11, Screenworks, Highbury Grove, Highbury and Islington, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided